CLINICAL TRIAL: NCT02007707
Title: A Family-Based Approach To Reduce Smoking in Vietnamese Men
Acronym: Tobacco LHW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TRDRP 22RT-0089
Record Dates: First submitted 2013-11-25; First posted 2013-12-11 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Tobacco Use Cessation; Healthy Eating
Keywords: Asian American; Vietnamese American; Smoking cessation; Community Health Worker; Lay Health Worker Outreach; Family Intervention
MeSH Terms: conditions — Tobacco Use Cessation; Smoking Cessation | interventions — Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tobacco LHW (Experimental): Quit Smoking For a Healthy Family - family-based psycho-education intervention using lay health worker (LHW) outreach.
  Interventions: Behavioral: Tobacco LHW
- Healthy Eating (Active Comparator): Eating Healthy and Physically Active for You and Your Family - This is a attention-control comparison group using a family-based psycho-education intervention delivered through lay health worker (LHW) outreach.
  Interventions: Behavioral: Healthy Eating

INTERVENTIONS:
Behavioral: Tobacco LHW — Quit Smoking For a Healthy Family - This is a family-based psycho-education intervention using lay health worker (LHW) outreach. LHW will be trained to recruit smoke-family dyads and provide education and information about tobacco and health, and smoking cessation resources through 2 small-group education sessions and 2 individual phone calls over a 2-month period.
  Arms: Tobacco LHW
Behavioral: Healthy Eating — Eating Healthy and Physically Active for You and Your Family - This is a attention-control comparison group using a family-based psycho-education intervention delivered through lay health worker (LHW) outreach. LHW will be trained to recruit smoke-family dyads and provide education and information about healthy eating and physical activity through 2 small-group education sessions and 2 individual phone calls over a 2-month period. Participants will receive writing information about smoking cessation resources.
  Arms: Healthy Eating

SUMMARY:
The goals of the study are to develop smoking cessation intervention using lay health worker (LHW) outreach and family involvement targeting Vietnamese Americans ages 18 and above in Santa Clara County, CA, to evaluate efficacy of the proposed intervention. The study is a two-arm randomized controlled trial targeting a total of 18 lay health workers (LHW) and 108 dyads of a smoker and a family member from the same household. The hypotheses are:

H. At 6-month post initiation of the intervention, Vietnamese male daily smokers who receive the proposed -Quit Smoking For a Healthy Family Intervention, a Family-based Intervention (FI), will be more likely to achieve biochemically verified 7-day point prevalence of smoking abstinence when compared to those receiving an attention control intervention (CI).

H2. At 6-month, FI participants we be more likely to report making at least one 24-hour quit attempt than those in CI.

H3. At 6-month, FI participants will be more likely to report using a recommended evidence-based smoking cessation resource (quitline, FDA-approved smoking cessation medications, advice from health professionals) than those in CI

ELIGIBILITY:
Inclusion Criteria:

* self-identified as Vietnamese, Vietnamese-American, or Vietnamese-Chinese;
* Vietnamese speaking;
* reside in the Santa Clara County, California
* plan to stay in the area (Santa Clara County, California) for the next 6 months
* for the smoker participants, they must be male and have smoked at least 1 cigarette daily in the past 7 days.
* for family member participants, the participant must live in the same household as the smoker participant to form a dyad.
* provide a valid contact telephone number for pre- and post-intervention assessments.

Exclusion Criteria:

- For smoker participants, currently engaging in assisted smoking cessation efforts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
smoking abstinence | 6-month
  biochemically verified 7-day point prevalence of smoking abstinence at 6-month post baseline (initiation of intervention)

SECONDARY OUTCOMES:
24-hour quit attempt | 6-month
  report making at least one 24-hour quit attempt at 6-month post baseline
resource utilization | 6-month
  report using a recommended evidence-based smoking cessation resource (quitline, FDA-approved smoking cessation medications, advice from health professionals) at 6-month post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Janice Y Tsoh, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Vietnamese Voluntary Foundation, San Jose, California
  - Immigrant Resettlement & Cultural Center (IRCC), Santa Clara, California